CLINICAL TRIAL: NCT00683033
Title: Contingency Management for Smoking in Substance Abusers
Acronym: R21
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UConn Health (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 08-081-2; R21DA021836-01A2 (NIH)
Record Dates: First submitted 2008-05-14; First posted 2008-05-23 (Estimated); Last update posted 2011-11-21 (Estimated); Status verified 2011-11

CONDITIONS: Cigarette Smoking
Keywords: Contingency Management; Cigarette Smoking Cessation; Substance Abusers
MeSH Terms: conditions — Cigarette Smoking; Tobacco Use Cessation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Brief counseling based on public health service guidelines.
  Interventions: Behavioral: Brief smoking cessation counseling
- B (Experimental): Brief counseling based on public health service guidelines for quitting smoking plus prize-based contingency management
  Interventions: Behavioral: Contingency Management; Behavioral: Brief smoking cessation counseling

INTERVENTIONS:
Behavioral: Contingency Management — For 4 weeks starting on the quit date, daily brief (about 5 minutes) counseling based on public health service guidelines for quitting smoking is delivered. Expired carbon monoxide (CO) tests are conducted twice daily and urinary cotinine tests are conducted once each week. Participants earn the opportunity to win prizes for submitting samples that meet smoking abstinence criteria (e.g., CO ≤ 6ppm; cotinine ≤ 30ng/mL).
  Arms: B
Behavioral: Brief smoking cessation counseling — For 4 weeks starting on the quit date, daily brief (about 5 minutes) counseling based on public health service guidelines for quitting smoking. Expired carbon monoxide tests are conducted twice daily and urinary cotinine tests are conducted once each week.

SUMMARY:
Patients (N=102) who meet diagnostic criteria for alcohol, cocaine, marijuana, or opiate abuse or dependence will meet with research staff on two days for quit preparation sessions (2 per day). These sessions include testing a breath sample for evidence of smoking twice each day (separated by at least 5 hours), counseling based on Public Health Service (PHS) guidelines for quitting smoking during the second session each day, and setting a quit date. After these sessions, participants will be randomly assigned to one of two 4-week conditions: (a) standard care or (b) standard care plus prize CM for smoking abstinence with the opportunity to win prizes for submitting samples that meet smoking abstinence criteria (e.g., CO ≤ 6ppm; cotinine ≤ 30ng/mL). Nicotine withdrawal and related measures will be assessed throughout the intervention. Follow-up data will be collected through 6-months post-quit date.

ELIGIBILITY:
Inclusion Criteria:

* current alcohol, cocaine, marijuana, or opiate abuse or dependence
* smoke ≥ 10 cigarettes per day
* expired CO > 8 ppm
* self-reported interest in quitting smoking,
* ≥ 18 years old
* willing to provide names, addresses and phone numbers of individuals to assist in locating the participant for follow-up evaluations,
* English speaking

Exclusion Criteria:

* currently receiving behavioral therapy or pharmacotherapy for smoking plan to use pharmacotherapy in this quit attempt
* serious, uncontrolled psychiatric illness (e.g., acute schizophrenia, suicide risk)
* cognitive impairment
* in recovery for pathological gambling

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2008-05; Primary Completion 2010-10 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
Cigarette smoking abstinence. | Daily through the 4-week intervention and at follow-up interviews 1, 2, 3, and 6 months following the quit date.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila M Alessi, Ph.D., Principal Investigator — UConn Health
Locations (1):
- University of Connecticut Health Center, Farmington, Connecticut, United States